CLINICAL TRIAL: NCT07399821
Title: A Phase Ib/II First-in-human Imaging Study of Anti-GD2-800CW in Patients With Neuroblastoma
Brief Title: An Imaging Study of Anti-GD2-800CW in Patients With Neuroblastoma
Acronym: GLOW-FISH
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Princess Maxima Center for Pediatric Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2023-507596-22-00; 2023-507596-22-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-27; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-11

CONDITIONS: Neuroblastoma
Keywords: Neuroblastoma; Fluorescence Guided Surgery; NIR fluorescence; pediatric oncology
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Intervention Model Description: Each subject will receive a single infusion of anti-GD2-800CW. There will be 3 different dose levels investigated in the GLOW-FISH trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-GD2-800CW (Experimental): Participants will receive a single dose of anti-GD2-800CW 96 hours prior to surgery.
  Interventions: Drug: anti-GD2-800CW

INTERVENTIONS:
Drug: anti-GD2-800CW — Participants will receive a single dose of anti-GD2-800CW 96 hours prior to surgery. In phase Ib, using a 3+3 design, a dose escalation is performed to determine the RP2D.

SUMMARY:
This is a non-randomized, open label phase Ib/II dose-escalation and expansion study designed to define the recommended dose of anti-GD2-800CW in pediatric neuroblastoma patients. The aim of this imaging study is to determine a safe and effective dose of anti-GD2-800CW for intra-operative detection of neuroblastoma using NIR fluorescence.

DETAILED DESCRIPTION:
Neuroblastoma is the most commonly diagnosed extracranial solid tumor in young children. It is a neural crest derived malignancy, which are the cells that give rise to the sympathetic nervous system, and can therefore be located in different body compartments. However, it occurs most frequently (80%) in the abdomen. Current treatment involves debulking surgery using standard-of-care, not assisted by intra-operative visualization of the tumor. In this current situation there is, i) a high risk of severe complications such as bleeding or unplanned nephrectomy (40%), ii) a high chance of >10% residual tumor tissue, and iii) difficulty distinguishing neuroblastoma subtypes with varying malignancy. Therefore, there is a high need for new tools enabling tumor-specific intra-operative visualization to assist the surgeon. This will reduce surgical complications and ensure neuroblastoma cells can be visualized and resected during surgery. Over the past years, Fluorescence Guided Surgery (FGS) has proven to be a useful intraoperative tool to increase the visibility of the tumor in various adult cancers. Our group has developed and validated a tumor-specific fluorescent agent, anti-GD2-800CW, that can be used to visualize neuroblastoma during surgery. Anti-GD2-800CW consists of two substances. Firstly, the monoclonal antibody anti-GD2, also known as Qarziba or Dinutuximab-beta, which binds to Disialoganglioside 2 (GD2), a tumor-associated antigen specifically expressed by neuroblastoma, most melanomas and several other tumors. Immunotherapy with anti-GD2 is now standard therapy for high-risk neuroblastoma treatment in patients aged 12 months and above. Secondly, the near-infrared (NIR) fluorescent dye, IRDye800CW, which is used extensively in clinical trials as fluorescent imaging agent without any known adverse events (AEs). The aim of this study is to investigate the safety and efficacy of this novel agent, anti-GD2-800CW, to visualize neuroblastoma during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with the diagnosis of neuroblastoma as defined by histopathology (confirmed by the PMC Department of Pathology), who will be operated for NB as standard of care procedure
* Patients older than 1 year of age and not older than 18 years.
* Written informed consent from patients and/or from parents or legal guardians, according to local law and regulations

Exclusion Criteria:

* Previous treatment with Dinutuximab-beta, either alone or in combination with chemotherapy
* Pregnancy or positive pregnancy test (urine or serum) in females of childbearing potential. Pregnancy test must be performed within during the screening period and before the administration of the IMP.
* Breast feeding.
* Sexually active participants not willing to use highly effective contraceptive method (pearl index <1) as defined in CTFG HMA 2020 (Appendix I) during trial participation and until 6 months after end of protocol therapy.
* Patients that received prior treatment with chimeric antibodies.

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 22 (Estimated)
Dates: Start 2025-11-05 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
To establish the recommended phase 2 dose (RP2D), based on efficacy and safety, of the anti-GD2-800CW fluorescent imaging agent in pediatric patients with neuroblastoma. | Through escalation phase completion, an average of 1 year.
  Establishing the recommended phase 2 dose (RP2D), based on efficacy and safety, of the anti-GD2-800CW fluorescent imaging agent.
To investigate safety of anti-GD2-800CW based on treatment related new AEs. | From IMP administration to 4 days after surgery
  Registration of new AEs.

SECONDARY OUTCOMES:
To assess the pharmacodynamic characteristics of an i.v. injection of anti-GD2-800CW. | From just before infusion to 4 days after surgery.
  Assessment will be done by measuring Anti Drug Antibody formation using an ADA binding assay. Blood samples will be taken at 8 time points.
To assess the pharmacokinetic characteristics of an i.v. injection of anti-GD2-800CW. | From just before infusion to 4 days after surgery.
  Assessment will be done by by measuring plasma levels Dinutuximab. Dinutuximab levels will be measured over time to create a concentration-time profile per patient. Blood samples will be taken at 8 time points.
To correlate clinical imaging data with histopathology data to determine the accuracy for depicting GD-2 expressing vital tumor cells. | From start surgery to 3 weeks after surgery when the PA results are analyzed.
  Pathologic status of removed fluorescent tissue and of removed fluorescent tissue will be compared to fluorescent status.
To assess the intra-operative usability of anti-GD2-800CW to distinguish tumor tissue from surrounding tissue on eyesight of the surgeons. | From start surgery to 3 weeks after surgery when the PA results are analyzed.
  Score of ≥ 4.0 on a Likert scale of 1-5 based on the judgement of three surgeons. They will grade the intra-operative visibility of the fluorescence and whether a clear distinction can be made on eyesight between tumor and surrounding tissue based on fluorescence.
To assess whether tumor load influences the fluorescence intensity. | From pre-operative scan to when PA results are analyzed, 3 weeks after surgery.
  Tumor load will be examined in preoperative imaging with the tumor volume (cm3). Additionally, we will denote the histopathological outcome with an estimation of vital tumor present after resection.

CONTACTS AND LOCATIONS:
Locations (1):
- Prinses Maxima Centrum, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No
Only IPD used in the results publication.